CLINICAL TRIAL: NCT02254070
Title: Influence of Different Degrees of Renal Impairment on the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of 1.0 mg of BIBT 986 BS Given as a Single Dose Infusion Over 30 Minutes in Subjects With Normal Renal Function and Patients With Different Degrees of Renal Impairment in an Open, Group Comparison Design
Brief Title: Influence of Different Degrees of Renal Impairment on the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of BIBT 986 BS in Subjects With Normal Renal Function and Patients With Different Degrees of Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1192.12
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy

ARMS (1):
- BIBT 986 BS (Experimental)
  Interventions: Drug: BIBT 986 BS

INTERVENTIONS:
Drug: BIBT 986 BS

SUMMARY:
To assess the influence of different degrees of renal impairment on safety, tolerability, pharmacodynamics and pharmacokinetics of 1.0 mg of BIBT 986 BS given as a single dose infusion over 30 minutes in comparison to a normal renal function

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects determined by results of screening with a creatinine clearance >80 mL/min (Group 1)
* Renally impaired male or female subjects determined by results of screening with the following creatinine clearance results:

  * creatinine clearance 51-80 mL/min (Group 2)
  * creatinine clearance 31-50 mL/min (Group 3)
  * creatinine clearance ≤ 30 mL/min (Group 4)
  * subjects requiring hemodialysis (Group 5)
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age >=18 and <=75 years
* BMI >=18.5 and <=29.9 kg/m2 for Groups 1+2
* BMI >=18.5 and <=32 kg/m2 for Groups 3, 4 and 5

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate, and electrocardiogram) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Relevant history of orthostatic hypotension, fainting spells or blackouts
* Abnormal PT, TT, aPTT (must be within the normal range after no more than one repeated test), thrombocytes < 150000/μl (two repeats of the first test)
* Evidence of haematuria either macroscopically detectable or microscopic on urinalysis (normal microscopic results after no ore than one repeated test)
* Evidence of blood dyscrasia, haemorrhagic diathesis, severe thrombocytopenia, cerebrovascular haemorrhage, bleeding tendencies associated with active ulceration or overt bleeding of gastrointestinal, respiratory or genitourinary tract or any disease or condition with haemorrhagic tendencies (e.g. cerebral aneurysm, dissecting aorta, CNS trauma, retinopathy, nephrolithiasis)
* Recent or contemplated diagnostic or therapeutic procedures with potential for uncontrollable bleeding (e.g. spinal puncture, lumbar block anaesthesia, surgery of central nervous system (CNS) or eye or surgery resulting in large open surfaces) within 14 days before or after drug administration of this clinical trial
* Occult blood in 1 of 3 subsequent faecal samples collected for the pre-study examination
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* For women with childbearing potential: no reliable contraception (accepted methods are intra uterine device, hormonal contraceptives, bilateral tubal ligation, hysterectomy, condoms) or pregnancy (known or detected by a positive pregnancy test) or breast feeding period
* Intake of drugs with a long half-life (> 24 hours) (< 1 month prior to administration or during the trial)
* Use of any drugs, within 14 days prior to administration or during the trial
* Participation in another trial with an investigational drug (< 2 months prior to administration or during trial)
* Smoker (> 10 cigarettes or >3 cigars or >3 pipes/day)
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation or loss > 400 ml, < 1 month prior to administration or during the trial
* Excessive physical activities < 5 days prior to administration of study drug or during trial
* Clinically relevant laboratory abnormalities
* Veins unsuited for i.v. puncture and administration of prolonged infusions on either arm (e.g. veins which are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture, etc.)

Renally impaired subjects (Group 2, 3, 4 and 5) who meet any of the following criteria will not be entered into this trial:

* Moderate and severe concurrent liver function impairment (e.g., due to hepatorenal syndrome)
* Gastrointestinal, respiratory, cardiovascular, metabolic, immunologic or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Relevant history of orthostatic hypotension, fainting spells or blackouts
* Abnormal values for PT, TT, aPTT and thrombocytes considered by the investigator or one of the co-investigators to be clinically relevant
* Hemoglobin concentration <9 mg/dl
* Evidence of blood dyscrasia, haemorrhagic diathesis, severe thrombocytopenia, cerebrovascular haemorrhage, bleeding tendencies associated with active ulceration or overt bleeding of gastrointestinal, respiratory or genitourinary tract or any disease or condition with haemorrhagic tendencies (e.g. cerebral aneurysm, dissecting aorta,CNS trauma, retinopathy, nephrolithiasis) considered by the investigator or one of the co-investigators to be clinically relevant
* Recent or contemplated diagnostic or therapeutic procedures with potential for uncontrollable bleeding (e.g. spinal puncture, lumbar block anaesthesia, surgery of CNS or eye or surgery resulting in large open surfaces) within 14 days before or after drug administration of this clinical trial
* Occult blood in 1 of 3 subsequent faecal samples collected for the pre-study examination
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* For women with childbearing potential: no reliable contraception (accepted methods are intra uterine device, hormonal contraceptives, bilateral tubal ligation, hysterectomy, condoms) or pregnancy (known or detected by a positive pregnancy test) or breast feeding period
* Faecal occult blood (FOB) in 1 of 3 subsequent samples collected for the pre-study examination
* Use of any drugs which have an influence on the blood clotting within 14 days prior to administration or during the trial (except heparin for hemodialysis patients)
* Participation in another trial with an investigational drug (< 2 months prior to administration or during trial)
* Smoker (> 10 cigarettes or >3 cigars or >3 pipes/day)
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation or loss > 400 ml, < 1 month prior to administration or during the trial
* Excessive physical activities < 5 days prior to administration of study drug or during trial
* Clinically relevant laboratory abnormalities
* Veins unsuited for i.v. puncture and administration of prolonged infusions on either arm (e.g. veins which are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2003-06; Primary Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Maximum measured concentration of the analyte in plasma (Cmax) | Up to 48 hours after drug administration
Time to reach the maximum concentration of the analyte in plasma (tmax) | Up to 48 hours after drug administration
Total area under the plasma drug concentration-time curve from time zero to infinity (AUC0-∞) | Up to 48 hours after drug administration
Area under the concentration-time curve of the analyte in plasma from zero time to the time of the last quantifiable drug concentration (AUC0-tz) | Up to 48 hours after drug administration
Terminal rate constant of the analyte in plasma (λz) | Up to 48 hours after drug administration
Terminal half-life of the analyte in plasma (t1/2) | Up to 48 hours after drug administration
Mean residence time of the analyte in the body after intravenous infusion (MRTinf) | Up to 48 hours after drug administration
Total clearance of the analyte from plasma following intravascular administration (CL) | Up to 48 hours after drug administration
Apparent volume of distribution at steady state following an intravascular dose (Vss) | Up to 48 hours after drug administration
Apparent volume of distribution during the terminal phase λz following an intravascular dose (Vz) | Up to 48 hours after drug administration
Amount of drug excreted in the urine (Ae) | Up to 48 hours after drug administration
Change in activated partial thromboplastin time (aPTT) | Up to 48 hours after drug administration
Change in ecarin clotting time (ECT) | Up to 48 hours after drug administration
Change in International Normalized Ratio (INR) | Up to 48 hours after drug administration
Change in thrombin time (TT) | Up to 48 hours after drug administration
Plasma concentration of the analyte at the end of the intravenous infusion (CT) | 29 minutes after drug administration
Number of participants with clinically significant changes in vital signs | Up to 3 days after drug administration
  Blood pressure and pulse rate
Number of participants with clinically significant changes in ECG (electrocardiogram) | Up to 3 days after drug administration
Number of participants with abnormal changes in clinical laboratory parameters | Up to 3 days after drug administration
Number of participants with adverse events | Up to 3 days after drug administration
Change in prothrombin time (PT) | Up to 48 hours after drug administration
partial area under the concentration time curve (from time 0 to last sampling time preceding hemodialysis in any of the patients) (AUCt1-t2) | Up to 48 hours after drug administration
fraction of administered drug excreted unchanged in urine over the respective time interval (fe) | Up to 48 hours after drug administration
Renal clearance of the analyte from plasma following intravascular administration (CLR) | Up to 48 hours after drug administration